CLINICAL TRIAL: NCT03456674
Title: Evaluation of the Lutronic LaseMD System for the Treatment of Melasma
Brief Title: LaseMD System for the Treatment of Melasma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CynosureLutronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L18002
Record Dates: First submitted 2018-02-26; First posted 2018-03-07 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Intervention Model Description: A single cohort of study subjects will receive study treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- LaseMD System (Experimental): Subjects will receive LaseMD System treatment(s) for treatment of melasma.
  Interventions: Device: LaseMD System

INTERVENTIONS:
Device: LaseMD System — A non-invasive fractional thulium laser delivering a wavelength of light energy as a fractionated array of microbeams to be absorbed by and damage the target molecule, a chromophore.

SUMMARY:
This study will evaluate the clinical outcomes associated with use of the LaseMD Laser System for the treatment of melasma.

DETAILED DESCRIPTION:
This clinical trial is a designed as a prospective, multi-site, non-randomized study of 20 subjects. Subjects will receive up to 5 study treatments completed 21 days apart. Phone follow-up will occur at Day 3 following each treatment for the assessment of adverse events and expected treatment effects. Post-treatment follow-up will be completed prior to the next subsequent treatment and at Days 30, 90 and 180 following the last treatment to assess adverse events and expected treatment effects, capture digital images, and assess efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Female, age 18 years and older.
2. Subject in good health.
3. Fitzpatrick Skin Type I to IV.
4. Moderate to severe melasma (Melasma Severity Scale, score 2 or 3).
5. Understands and accepts the obligation not to undergo any other procedures in the areas to be treated through the follow-up period.
6. Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
7. Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study.
8. Absence of physical or psychological conditions unacceptable to the investigator.
9. Willingness and ability to provide written consent for study-required photography and adherence to photography procedures (i.e., removal of jewelry and makeup).
10. Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure.

Exclusion Criteria:

1. Inability to understand the protocol or to give informed consent.
2. Presence of an active systemic or local skin disease that may affect wound healing.
3. History of keloids or poor wound healing.
4. Significant scarring in the area(s) to be treated that would interfere with assessing results.
5. Open wounds or lesions in the area(s) to be treated.
6. Excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin in the area(s) to be treated.
7. History of chronic drug or alcohol abuse.
8. History of collagen vascular disease.
9. History of autoimmune disease.
10. Subjects with sensitivity or allergy to pre-treatment medication, EMLA Cream (Lidocaine/Prilocaine).
11. Subjects with sensitivity or allergy to post-treatment cosmeceuticals, Tranexamic Acid and/or coconut.
12. Subjects with photosensitive skin.
13. Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
14. Subjects who are pregnant or lactating or anticipate becoming pregnant during the study.
15. Subjects who anticipate the need for inpatient surgery or overnight hospitalization during the study.
16. Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
17. Concurrent enrollment in any study involving the use of investigational devices or drugs.
18. Current smoker or history of smoking in the last five years.
19. Current user of any nicotine-containing products, e.g., e-cigarettes, Nicorette gum, nicotine patches, etc.
20. Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
21. History of surgical or cosmetic treatments in the area(s) to be treated within the past 6 months.
22. Microdermabrasion, or prescription level glycolic acid treatment to the treatment area(s) within 4 weeks prior to study participation or during the study.
23. History of hormone treatment, such as estrogen, progesterone and/or oral contraceptives, initiated within 3 months of study participation, or planning to discontinue hormone therapy during the study, as applicable.
24. Use of any prescription skin-lightening agent (such as tranexamic acid or hydroquinone), isotretinoin (or other retinoid), photo-sensitizing medication, or corticosteroid within 6 months of and during study participation.
25. History or current use of the following prescription medications:

    1. Accutane or other systemic retinoids within the past twelve months;
    2. Topical Retinoids within the past two weeks; and/or
    3. Antiplatelet agents/Anticoagulants (Coumadin, Heparin, Plavix) within the past two weeks.
    4. Psychiatric drugs that in the investigators opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-02-07 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in the Melasma Area and Severity Index (MASI) from Baseline | From baseline to 30 Days following the last study treatment.
  A change in MASI score from baseline to post-treatment. The MASI quantifies the pigmentation area, darkness, and homogeneity, assessing four areas of the face for hyperpigmentation: forehead, right malar region, left malar region and chin, corresponding to 30%, 30%, 30% and 10% of the total face. The melasma area in each region is given a numeric value from 1 (<10%) to 6 (90-100%) in each of the four regions. Darkness of pigment is compared to normal skin in each area on a scale of 0 (absent) to 4 (severe). Homogeneity is based on a scale of 0 (minimal) to 4 (maximal). The MASI score is then calculated as the sum of severity rating of darkness and homogeneity, multiplied by the value of area involved. The maximum score is 48; the minimum score is 0.

SECONDARY OUTCOMES:
Improvement in the Melasma Area and Severity Index (MASI) from Baseline | From baseline to Days 90 and 180 following the last study treatment.
  A change in MASI score from baseline to post-treatment. The MASI quantifies the pigmentation area, darkness, and homogeneity, assessing four areas of the face for hyperpigmentation: forehead, right malar region, left malar region and chin, corresponding to 30%, 30%, 30% and 10% of the total face. The melasma area in each region is given a numeric value from 1 (<10%) to 6 (90-100%) in each of the four regions. Darkness of pigment is compared to normal skin in each area on a scale of 0 (absent) to 4 (severe). Homogeneity is based on a scale of 0 (minimal) to 4 (maximal). The MASI score is then calculated as the sum of severity rating of darkness and homogeneity, multiplied by the value of area involved. The maximum score is 48; the minimum score is 0.
Clinician assessment of overall aesthetic improvement. | From baseline to Days 30, 90 and 180 following last treatment.
  Overall aesthetic improvement based on completion of a 5-point Clinician Global Aesthetic Improvement Scale, based on a live assessment of the subject while comparing to the subject's pre-treatment photographs, and based on a comparison of the subject's pre-treatment photographs to the current post-treatment photograph. Aesthetic improvement will be based on the following definitions:
  1. = Very Much Improved: Optimal cosmetic result.
  2. = Much Improved: Marked improvement in appearance from the initial condition, but not completely optimal.
  3. = Improved: Obvious improvement in appearance from initial condition
  4. = No Change: The appearance is essentially the same as the original condition.
  5. = Worse: The appearance is worse than the original condition.
Subject assessment of overall aesthetic improvement. | From baseline to Days 30, 90 and 180 following last treatment.
  Overall aesthetic improvement based on completion of a 5-point Subject Global Aesthetic Improvement Scale. Subjects will complete the scale based on a live assessment referring to a hand mirror and their pre-treatment photographs, and based on a comparison of their pre-treatment photographs to the current post-treatment photograph. Aesthetic improvement will be based on the following definitions:
  1. = Very Much Improved: Optimal cosmetic result.
  2. = Much Improved: Marked improvement in appearance from the initial condition, but not completely optimal.
  3. = Improved: Obvious improvement in appearance from initial condition
  4. = No Change: The appearance is essentially the same as the original condition.
  5. = Worse: The appearance is worse than the original condition.
Improvement in the Melasma Quality of Life Scale (MELASQOL) from baseline | From baseline to Day 30 following last treatment.
  The Melasma Quality of Life Scale assesses the effect melasma has on the quality of life of sufferers on a scale of 1 (not bothered at all) to 7 (bothered all of the time), rating the following questions:
  1. The appearance of your skin condition
  2. Frustration about your skin condition.
  3. Embarrassment about your skin condition.
  4. Feeling depressed about your skin condition.
  5. The effects of your skin condition on your interactions with other people.
  6. The effects of your skin condition on your desire to be with people.
  7. Your skin condition making it hard to show affection.
  8. Skin discoloration making you feel unattractive to others.
  9. Skin discoloration making you feel less vital or productive.
  10. Skin discoloration affecting your sense of freedom.
Patient Satisfaction Questionnaire | Day 30 following last treatment.
  Patient satisfaction will be evaluated based on subjects' completion of a patient satisfaction questionnaire while referring to a hand mirror and their pre-treatment photographs and their Day 30 follow-up photographs. Subjects will be asked to document Yes/No as to whether they notice any improvement in how the melasma on their face looks; beyond changes to the melasma pigment specify any changes they see in the treated areas, e.g., skin texture improvement, skin tone improvement, fine lines and wrinkles improvement, etc.; characterize their level of satisfaction with study treatment based on 5 levels of satisfaction: Very satisfied, Satisfied, Slightly Satisfied, Neither Satisfied or Dissatisfied, Dissatisfied; document Yes/No if they would recommend the treatment to friends and family members.
Treatment-related pain | For the duration of each study treatment
  During study treatments, subjects' pain levels will be monitored using a validated Numeric Rating Scale (0-10), with 0 being 'No Pain' and 10 being the 'Worst Possible Pain'.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Larson, MBA, Study Director — Sponsor GmbH
Locations (1):
- Laser and Skin Surgery Center of New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No